CLINICAL TRIAL: NCT05760196
Title: A Prospective, Multicenter, High- and Low-dose Radiotherapy Combined With PD-1 Inhibitors and GM-CSF in the Treatment of Advanced Recurrent Metastatic Head and Neck Tumors
Brief Title: Radiotherapy Combined With PD-1 Inhibitor and GM-CSF for Advanced Recurrent Metastatic Head and Neck Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiangpan Li (Other)
Responsible Party: Sponsor-Investigator, Xiangpan Li, Professor, Renmin Hospital of Wuhan University
Organization: Renmin Hospital of Wuhan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WDRY2022-K266
Record Dates: First submitted 2023-02-25; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Objective Response Rate
MeSH Terms: interventions — Granulocyte-Macrophage Colony-Stimulating Factor; spartalizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recurrent or metastatic advanced head and neck malignancy (Experimental): Patients with a clear pathological diagnosis, imaging diagnosis, and history, no clear recommended standard treatment or inability to tolerate standard treatment, and a clear measurable lesion
  Interventions: Drug: GM-CSF

INTERVENTIONS:
Drug: GM-CSF — PD1 antibody is held every three weeks, and GM-CSF is used once every three weeks on days 1-14. Until the patient progresses disease or intolerable toxicity.
  Other Names: PD-1 antibody

SUMMARY:
This is an intervention study, aiming to use high and low dose radiotherapy combined with PD-1/PD-L1 inhibitor combined with GM-CSF to observe the effect of anti-tumor immunity and long-term therapeutic response rate, and to explore a new treatment model for patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. Patients with recurrent or metastatic advanced head and neck malignancies (including nasopharyngeal malignancies), with a clear pathological diagnosis, imaging diagnosis, and medical history, no clearly recommended standard treatment regimen or inability to tolerate standard treatment regimens, and clear measurable lesions (>1 cm);
3. Patients with squamous cell carcinoma who progress after first-line antineoplastic therapy must include a platinum-containing combination chemotherapy or platinum-based concurrent chemoradiotherapy, and patients with secondary resistance after previous anti-PD-1/L1 therapy may also be enrolled;
4. There is no standard regimen recommended by guidelines after first-line treatment failure in patients with non-squamous cell carcinoma (eg, adenoid cystadenocarcinoma, lung metastases, sarcoma, etc.);
5. At least one lesion with a diameter of 1 cm to 5 cm (metastases ≥1 cm, if the patient has large metastases, partial tumor irradiation can be allowed) can be treated with radiation therapy at 16 to 24 Gy/2-3Fx doses; Lymph nodes can be used as stand-alone measurable lesions (if lymph nodes are evaluated as an evaluation lesion, they must meet the criteria for target lesions, see RECIST1.1 for definition of a lymph node target lesion);
6. Patients who have previously received radical radiotherapy need to have an interval of more than 6 months; Patients with an interval of more than 6 months from the previous radiotherapy;
7. In the past 6 months, there has been no acute coronary syndrome or malignant arrhythmia;
8. ECOG (Eastern Cooperative Oncology Group), score 0-2, life expectancy assessment ≥ 3 months;
9. There were no previous severe hematopoietic, cardiac, pulmonary, hepatic, or renal dysfunction or immunodeficiency;
10. Ejection fraction of cardiac color Doppler ultrasound ≥ 50%;
11. Myocardial enzyme profile and NT-proBNP do not exceed twice the upper limit of normal;
12. Troponin and CKMB values do not exceed twice the normal upper limit;
13. Patients who have had grade 2 or higher AV block in the past six months and need to consider pacemakers will not be included;
14. Blood pressure hypertension≤ 160mmHg and/or low pressure≤90mmHg. 1 week prior to enrollment, the level of organ function meets the following criteria:

    Bone marrow function: hemoglobin ≥ 80g/L, white blood cell count ≥ 3.5*10^9/L or neutrophil count ≥1.5*10^9/L, platelet count ≥ 100*10^9/L, CD8+ T lymphocyte absolute value ≥200/μL; Liver: serum total bilirubin level ≤ 1.5 times the upper limit of normal, when the serum total bilirubin level > 1.5 times the upper limit of normal, direct bilirubin level must ≤ the upper limit of normal, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times the upper limit of normal; (5.0 times ≤the upper limit of normal in patients with liver metastases); Kidney: serum creatinine level < 1.5 times the upper limit of normal or creatinine clearance ≥ 50ml/min, urea nitrogen ≤ 200mg/L; serum albumin≥ 30g/L;
15. Patients must have the ability to understand and voluntarily sign informed consent forms.

Exclusion Criteria:

1. Exclude single shot oligo transfer;
2. Pregnant or breastfeeding women;
3. Those who have a history of other malignant diseases in the past 5 years, except for cured skin cancer and cervical carcinoma in situ;
4. Patients with a history of uncontrolled epilepsy, central nervous system disease, or psychiatric disorders, as judged by the investigator, may hinder the signing of informed consent or affect the patient's adherence to drug therapy;
5. Clinically severe (i.e., active) heart disease such as symptomatic coronary heart disease, New York Heart Association (NYHA) class II or more congestive heart failure or severe arrhythmias requiring pharmacological intervention, or a history of myocardial infarction within the last 12 months;
6. Organ transplantation requires immunosuppressive therapy;
7. Known major active infection, or major blood, kidney, metabolic, gastrointestinal, endocrine function or metabolic disorders, or other serious uncontrolled concomitant diseases. Those who are allergic to any of the ingredients used in the study;
8. Those with a history of immunodeficiency, including those who test positive for HIV or have other acquired or congenital immunodeficiency disorders, or have a history of organ transplantation, or who have other immune-related disorders that require long-term oral hormone therapy;
9. Are in the period of acute and chronic TB infection (positive T-spot test, chest x-ray in patients with suspected tuberculosis);
10. Other circumstances that the investigator does not consider suitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 36 months
  Objective tumor response, including CR and PR, was assessed using RECIST version 1.1.

SECONDARY OUTCOMES:
Toxic reaction | 36 months
  Guidelines for Toxicity Management of CTC 5.0 Standard CSCO ESMO irAE.
Overall survival | 36 months
  The time between enrolment in the study and death from any cause.
Duration of remission | 36 months
  The time from the first confirmed CR or PR to the first occurrence of PD, or to death if it occurs during treatment.
Disease control rate | 36 months
  Refers to the percentage of cases with CR, PR, and SD (≥4 weeks) in patients with evaluable efficacy.
Progression-free survival | 36 months
  The time between initial use of the investigational drug and tumor progression/recurrence or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Xiangpan Li, Principal Investigator — Renmin Hospital of Wuhan University
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China